CLINICAL TRIAL: NCT06986564
Title: Agreement Between Multidisciplinary Cancer Board Decisions and ChatGPT-4O in Clinical Decision-Making: A Cross-Sectional Observational Study
Brief Title: Evaluation of Decision Compatibility Between a Multidisciplinary Cancer Board and ChatGPT-4O
Status: Completed | Type: Observational
Sponsor: Sebahattin Celik MD (Other)
Responsible Party: Sponsor-Investigator, Sebahattin Celik MD, Professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Other Study IDs: 2024-050695
Record Dates: First submitted 2024-12-20; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Artificial Intelligence
Keywords: Clinical decision agreement study; Cancer; Artificial intelligence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the decisions of a multidisciplinary cancer board at Van research and educational Hospital with those generated by ChatGPT-4O. Patient data, including age, gender, comorbidities, clinical findings, laboratory results, radiology, and pathology reports, will be collected and recorded in patient files. These records will then be converted into a textual format appropriate for input into the ChatGPT-4O model. Statistical analyses will be conducted to assess the level of agreement between the board's decisions and those of ChatGPT-4O, providing insights into their compatibility and potential utility in clinical practice.

DETAILED DESCRIPTION:
This study aims to evaluate the agreement between decisions made by a multidisciplinary cancer board at Van Hospital and those generated by the ChatGPT-4O model.

A total of 100 cancer patients presented to the multidisciplinary cancer board will be included in the study. Patient data, including age, gender, comorbidities, clinical findings, laboratory results, radiology, and pathology reports, will be systematically recorded and reformatted into text suitable for the ChatGPT-4O model. The AI model's decisions will then be compared to those made by the cancer board. Statistical analyses will be performed to quantify the level of agreement between the two decision sources.

The findings will provide insights into the compatibility between human-led multidisciplinary decisions and AI-driven recommendations, highlighting areas of agreement and disagreement.

This study will assess the potential utility of ChatGPT-4O in clinical oncology decision-making and explore whether AI models can support or complement traditional cancer board processes.

ELIGIBILITY:
Inclusion Criteria:

* above 18 y/o
* patients diagnosed with malignancy

Exclusion Criteria:

* patients who refused to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 cancer patients presented to the multidisciplinary cancer board will be included in the study. Patient data, including age, gender, comorbidities, clinical findings, laboratory results, radiology, and pathology reports, will be systematically recorded and reformatted into text suitable for the ChatGPT-4O model. The AI model's decisions will then be compared to those made by the cancer board. Statistical analyses will be performed to quantify the level of agreement between the two decision sources.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the agreement between decisions made by a multidisciplinary cancer board and those generated by the ChatGPT-4O model using kappa statistics. | 4 month
  Within the scope of this research, we aimed to elucidate the compatibility of artificial intelligence with the decisions made in patients brought to the multidisciplinary tumor council. We sought to answer whether we can accept artificial intelligence as a new member, other than humans, as a decision-support tool in the council.

CONTACTS AND LOCATIONS:
Overall Officials: Sebahattin Çelik, professor, Study Director — General surgery department chief
Locations (1):
- Van state hospital, general surgery department, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP